CLINICAL TRIAL: NCT01350037
Title: Alfentanil vs Remifentanil in Patient-controlled Sedation During ERCP.A Randomized Double-blind Study
Brief Title: Alfentanil Versus Remifentanil in Patient-controlled Sedation During Endoscopic Retrograde Cholangiopancreatography (ERCP)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maxim Mazanikov, M.D., Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: a002c; 2009-012398-36 (EudraCT Number)
Record Dates: First submitted 2011-05-05; First posted 2011-05-09 (Estimated); Last update posted 2012-07-06 (Estimated); Status verified 2012-07

CONDITIONS: Biliary Tract Diseases; Pancreatic Diseases
Keywords: patient-controlled sedation; propofol; alfentanil; remifentanil; endoscopic retrograde cholangiopancreatography
MeSH Terms: conditions — Biliary Tract Diseases; Pancreatic Diseases | interventions — Alfentanil; Remifentanil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- remifentanil (Active Comparator): sedative mixture for PCS consisting of propofol 10mg/ml 20 ml and remifentanil 50 mkg/ml 5 ml
  Interventions: Drug: remifentanil
- alfentanil 0.04 mg/ml (Active Comparator): sedative mixture for PCS consisting of propofol10 mg/ml 20 ml,alfentanil 0.5 mg/ml 2 ml, NaCL 9 mg/ml 3 ml
  Interventions: Drug: alfentanil
- alfentanil 0.08 mg/ml (Active Comparator): sedative mixture for PCS consisting of propofol 10 mg/ml 20 ml, alfentanil 0.5 mg/ml 4 ml,NaCl 9mg/ml 1ml
  Interventions: Drug: alfentanil

INTERVENTIONS:
Drug: alfentanil — Alfentanil is a potent but short-acting synthetic opioid analgesic drug, used for anaesthesia in surgery. It is an analogue of fentanyl with around 1/10 the potency of fentanyl and around 1/3 of the duration of action, but with an onset of effects 4x faster than fentanyl.It is an OP3 mu-agonist.Alfentanil is administered by the parenteral (injected) route for fast onset of effects and precise control of dosage.
  Other Names: Rapifen; Alfenta
  Arms: alfentanil 0.04 mg/ml; alfentanil 0.08 mg/ml
Drug: remifentanil — Remifentanil is a potent ultra short-acting synthetic opioid analgesic drug. It is given to patients during surgery to relieve pain and as an adjunct to an anaesthetic. Remifentanil is used for sedation as well as combined with other medications for use in general anesthesia. The use of remifentanil has made possible the use of high dose opioid and low dose hypnotic anesthesia, due to synergism between remifentanil and various hypnotic drugs and volatile anesthetics.It is administered in the form remifentanil hydrochloride and in adults is given as an intravenous infusion in doses ranging from 0.1 microgram per kilogram per minute to 0.5 (µg/kg)/min.
  Other Names: Ultiva
  Arms: remifentanil

SUMMARY:
Self-administration of propofol and opioid mixture by the patient him- or herself (patient-controlled sedation, PCS) could be successful alternative to the anesthesiologists-managed deep sedation during endoscopic retrograde cholangiopancreatography (ERCP). However, it is not known which opioid would be the most suitable for PCS. The aim of this double-blind study was to compare remifentanil and alfentanil in PCS during ERCP.

DETAILED DESCRIPTION:
Deep sedation with propofol has been suggested necessary for successful performance of endoscopic retrograde cholangiopancreatography (ERCP).Airway obstruction, hypoventilation and hypoxemia occurs in deeply sedated patients with a high incidence of 12-30%.As a result of frequent hypoxemia events, deep sedation is associated with increased morbidity and mortality.Careful monitoring of vital signs and involving of anesthesia-trained personal are recommended for deeply sedated patients.Self-administration of propofol by the patient him- or herself (patient-controlled sedation, PCS)could be a safer way to use propofol without the presence of an anesthesiologist. In comparison to the anesthesiologists managed deep sedation the main advantages of PCS are reduced consumption of anesthetics and faster recovery.A combination of propofol and different opioids is widely used for PCS however, it is not known which opioid would be the most suitable one. Remifentanil is a potent opioid with ultra short duration of action and usually administered as a constant infusion. The elimination half-life of alfentanil is 8-32 minutes being about 3 times longer, than that of remifentanil. Both opioids have been evaluated previously in PCS but comparative studies are lacking. This study was carried out in order to compare remifentanil and alfentanil in PCS during ERCP in terms of propofol consumption, sedation levels, endoscopist´s and patient's satisfaction. The investigators also sought information about frequency of sedation related complications associated with the different opioids.

ELIGIBILITY:
Inclusion Criteria:

* elective ERCP patients

Exclusion Criteria:

* allergy to propofol or opioid analgesics, drug addiction, inability to co-operate, ASA class greater than 3, or patient's refusal.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
consumption of propofol and opioid | one day
vital signs | one day
  Heart rate (HR), electrocardiogram (ECG), breathing rate, peripheral oxygen saturation (SpO2), end tidal carbon dioxide (EtCO2) constant monitoring. Noninvasive blood pressure (NIBP)measuring at 5 min intervals.

SECONDARY OUTCOMES:
sedation levels | one day
  Modified Observer's Assessment of Alertness and Sedation (MOAA/S) score
pain intensity | one day
  Numeric range scale
patient´s and endoscopist´s satisfaction with sedation | one day
incidence of nausea | one day

CONTACTS AND LOCATIONS:
Overall Officials: Reino Pöyhiä, MD,PhD, Study Director — Helsinki University Central Hospital, Department of Anesthesiology and Intensive Care; Maxim Mazanikov, MD, Principal Investigator — Helsinki University Central Hospital,Department of Anesthesiology and Intensive Care; Martti Färkkilä, MD,Professor, Principal Investigator — Helsinki University Central Hospital,Department of Medicine, Division of Gastroenterology; Leena Kylänpää, MD,PhD, Principal Investigator — Helsinki University Central Hospital,Department of Gastrointestinal and General Surgery; Jorma Halttunen, MD,PhD, Principal Investigator — Helsinki University Central Hospital,Department of Gastrointestinal and General Surgery; Outi Lindström, MD,PhD, Principal Investigator — Helsinki University Central Hospital,Department of Gastrointestinal and General Surgery; Harri Mustonen, DSc, Principal Investigator — Helsinki University Central Hospital, Department of Surgery; Marianne Udd, MD,PhD, Principal Investigator — Helsinki University Central Hospital,Department of Gastrointestinal and General Surgery
Locations (1):
- Helsiki University Central Hospital,Meilahti Hospital,Endoscopy unit, Helsinki, Uusimaa, Finland